CLINICAL TRIAL: NCT01750229
Title: Randomized Controlled Double-blind Cross-over Trial Evaluating the Role of Frequencies on Spinal Cord Stimulation in the Management of Failed Back Surgery Syndrome (SCS Frequency Study)
Brief Title: Spinal Cord Stimulation Frequency Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MedtronicNeuro (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1668
Record Dates: First submitted 2012-11-19; First posted 2012-12-17 (Estimated); Results first posted 2017-12-18 (Actual); Last update posted 2017-12-18 (Actual); Status verified 2017-05

CONDITIONS: Failed Back Surgery Syndrome
MeSH Terms: conditions — Failed Back Surgery Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- Sham (Sham Comparator): Frequency Setting - Sham
  Interventions: Device: Sham
- 1200 Hz (Experimental): Frequency Setting - 1200 Hz
  Interventions: Device: 1200 Hz
- 3030 Hz (Experimental): Frequency Setting - 3030 Hz
  Interventions: Device: 3030 Hz
- 5882 Hz (Experimental): Frequency Setting - 5882 Hz
  Interventions: Device: 5882 Hz

INTERVENTIONS:
Device: Sham — Frequency Setting - Sham
  Arms: Sham
Device: 1200 Hz — Frequency Setting - 1200 Hz
  Arms: 1200 Hz
Device: 3030 Hz — Frequency Setting - 3030 Hz
  Arms: 3030 Hz
Device: 5882 Hz — Frequency Setting - 5882 Hz
  Arms: 5882 Hz

SUMMARY:
The purpose of this study is to evaluate the role of frequency settings on spinal cord stimulation in the management of Failed Back Surgery Syndrome (SCS Frequency Study).

DETAILED DESCRIPTION:
Prospective, single-center, double-blinded, randomized crossover of 4 different stimulation frequencies: sham, 1200 Hz, 3030 Hz, and 5882 Hz.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old at the time of informed consent
* Willing and able to provide a signed and dated informed consent
* Capable of comprehending and consenting in English
* Willing and able to comply with all study procedures, study visits, and be available for the duration of the study
* On a stable dose (no new, discontinued or changes in) of all prescribed pain medications and willing/able to maintain or only decrease the dose of all prescribed pain medications
* Tried appropriate conventional medical management for their pain
* Not indicated for additional surgical treatment in the opinion of the referring physician or spinal surgeon
* Undergone previous spinal surgery
* Diagnosed with FBSS with appropriate pain score
* Primary pain at appropriate spinal level

Exclusion Criteria:

* Has an active implanted device, whether turned on or off
* Displays current signs of a systemic infection
* Pregnant or lactating, inadequate birth control, or the possibility of pregnancy during the study
* Has untreated major psychiatric comorbidity
* Has serious drug-related behavioral issues
* Has neurological abnormalities unrelated to Failed Back Surgery Syndrome
* Diagnosed with Raynaud disease
* Diagnosed with Fibromyalgia
* Has any active malignancy or has been diagnosed with cancer and has not been in remission for at least 1 year prior to screening
* Has secondary gains which, in the opinion of the investigator, are likely to interfere with the study
* Participating or planning to participate in another clinical trial
* Has characteristics/limits of household or close contacts involved in study (eg, family member already a study participant where blind could be broken)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2012-12; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adnan Al-Kaisy, Dr., Principal Investigator — Guy's and St Thomas' NHS Foundation Trust
Locations (1):
- Guy's and St. Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] O'Connell NE, Ferraro MC, Gibson W, Rice AS, Vase L, Coyle D, Eccleston C. Implanted spinal neuromodulation interventions for chronic pain in adults. Cochrane Database Syst Rev. 2021 Dec 2;12(12):CD013756. doi: 10.1002/14651858.CD013756.pub2. PMID 34854473

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 53 subjects were recruited between January 2013 and April 2015.
Pre-assignment Details: A total of 23 subjects discontinued prior to randomization due to eligibility criteria not met or withdrawal from the study.
Groups:
- All Randomized Subjects: Randomized phase subjects received all four frequency settings (Sham, 1200 Hz, 3030 Hz, and 5882 Hz), each for 3 weeks, in a randomized order.
Period: Randomized Crossover Phase
Arm/Group | All Randomized Subjects
Started | 30
Subject Received Sham | 24
Subjects Received 1200 Hz | 24
Subjects Received 3030 Hz | 24
Subjects Received 5882 Hz | 24
Protocol Violation | 4
Completed | 28
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1
Period: Long-term Follow-up Phase
Arm/Group | All Randomized Subjects
Started | 28 (Four subjects who had protocol violations continued to be followed in long-term follow-up phase.)
Completed | 25
Not Completed | 3
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Randomized Phase Subjects: Randomized phase subjects received all four frequency settings (Sham, 1200 Hz, 3030 Hz, and 5882 Hz), each for 3 weeks, in a randomized order.
Arm/Group | Randomized Phase Subjects
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.9 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 16
Region of Enrollment [Number; unit: participants]
  United Kingdom | 24
Baseline VAS back pain score [Mean (Standard Deviation); unit: units on a scale] — Visual Analog Scale (VAS) back pain scores were recorded once a day on a multi-day diary, where subjects rate the pain by making a vertical slash mark through the 0-10cm line that best describes their pain during the last 24 hours, with 0 = No pain and 10 = Worst pain imaginable. The higher VAS back pain score represented worse back pain. The average VAS back pain scores from 7 days in the diary were used for summary.
  units on a scale | 7.75 (1.13)

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale (VAS) on Back Pain
Description: Visual Analog Scale (VAS) back pain scores were recorded once a day on a multi-day diary, where subjects rate the pain by making a vertical slash mark through the 0-10cm line that best describes their pain during the last 24 hours, with 0 = No pain and 10 = Worst pain imaginable. The higher VAS back pain score represented worse back pain. The average VAS back pain scores from the last three days of diary prior to the follow-up visits were used for analysis.
Time Frame: 12 weeks
Population: Per-protocol population, subjects who followed the protocol and provided data for all four randomized crossover period were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Sham; 1200 Hz; 3030 Hz; 5882 Hz: Randomized phase subjects received all four frequency settings (Sham, 1200 Hz, 3030 Hz, and 5882 Hz), each for 3 weeks, in a randomized order.
Arm/Group | Sham | 1200 Hz | 3030 Hz | 5882 Hz
Number analyzed (Participants) | 24 | 24 | 24 | 24
units on a scale | 4.83 (2.45) | 4.51 (1.87) | 4.57 (2.09) | 3.22 (1.98)
Statistical Analysis 1: Comparison: Sham vs 1200 Hz vs 3030 Hz vs 5882 Hz; Test type: Superiority; p = 0.002, Mixed Models Analysis; Variables included in the Mixed Model were: baseline VAS back pain score, treatment group, and period

ADVERSE EVENTS:
Time Frame: Randomized crossover phase of 12 weeks
Arm/Group | Sham | 1200 Hz | 3030 Hz | 5882 Hz
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 1/24 | 0/24 | 1/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 2/24 | 0/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sham (N=24) | 1200 Hz (N=24) | 3030 Hz (N=24) | 5882 Hz (N=24)
Implant site pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sham (N=24) | 1200 Hz (N=24) | 3030 Hz (N=24) | 5882 Hz (N=24)
Implant site pain (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Trust and/or the PI may prepare the data derived from the study for publication. Data will be submitted to the Sponsor for review and comment prior to publication and at least sixty (60) days prior to submission for publication, public dissemination, or review by a publication committee.

All reasonable comments made by the Sponsor in relation to a proposed publication will be incorporated by the Trust and/or the Investigator into the publication.